CLINICAL TRIAL: NCT02839538
Title: A Comparative Randomised Study of the Analgesic Effect of Local Infiltration or Spinal Block for Haemorrhoidectomy
Brief Title: Comparative Study of the Analgesic Effect of Spinal Anesthesia or Infiltration Anesthesia for Hemorrhoidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luis Antonio Borges, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 37140514.9.000.5505
Record Dates: First submitted 2016-07-06; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Postoperative Pain
Keywords: infiltration; hemorrhoidectomy; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Local; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local Infiltration (Active Comparator): Induction of General Anesthesia with Propofol(2mg/Kg) and Atracurium(0,5mg/Kg) . Pulmonary ventilation with laryngeal mask and Propofol infusion ( 100mcg/Kg/min.) After , Infiltration of 0.75% ropivacaine (10 ml) each side block injection of local anesthetic at perianal.
  If necessary, fentanyl endovenous injection (50 mcg).
  Interventions: Procedure: Local Infiltration
- Subarachnoidal block (Other): Sedation with midazolam 2 mg. After , Spinal block with 10 mg of hyperbaric 0.5% bupivacaine. Injection of anesthetic at subarachnoidal space with Quincke needle 27G.
  If pain, local infiltration with lidocaine 1% (5 ml) in wound.
  Interventions: Procedure: Subarachnoidal block

INTERVENTIONS:
Procedure: Local Infiltration — Injection at perianal region with ropivacaine 0.75%(20ml)
  Other Names: local anesthesia
  Arms: local Infiltration
Procedure: Subarachnoidal block — Injection at subarachnoidal space with bupivacaine 0.5% ( 2ml)
  Other Names: spinal anesthesia
  Arms: Subarachnoidal block

SUMMARY:
Background and Objectives: Postoperative analgesia and early recovery are relevant for hospital discharge after hemorrhoidectomy. This study investigated the postoperative analgesic effect with local infiltration compared with spinal block.

Methods: This randomized study included 40 patients aged 18 to 60 years old. Local group (LG) received local infiltration under general anaesthesia; spinal group (SG) received a subarachnoid block. LG received general anaesthesia with propofol, atracurium and propofol infusion as well as a local infiltration of 20 ml 0.75% ropivacaine. SG received 2 ml of 0.5% hyperbaric bupivacaine. Analgesic supplementation was with 50µg of fentanyl for LG and 1% lidocaine for SG. There were assessed: postoperative pain intensity, sphincter relaxation, motor blockade of lower limbs, time to discharge, analgesic dose over 1 week and adverse effects.

DETAILED DESCRIPTION:
This is a prospective, randomized study, including 40 patients between 18 and 60 years, of both genders, ASA 1 or 2.

Patients in group 1( n= 19 ) will be submitted to spinal block and group 2 (n=21) to local infiltration. The spinal block will be performed with 10 mg of 0.5% bupivacaine. The infiltration will be performed with 10 ml of 0.75% ropivacaine on each side.

Will be evaluated: intensity of pain on a numerical scale from 0 to 10 every 30 minutes, relaxation of the sphincter muscles, intensity of pain after the operation every 30 minutes until reached the criteria for discharge, motor blocked of the lower limbs every 30 minutes, BP, HR, SO2, FR, other items that determine the conditions of discharge (urine output, nausea and vomiting), time to hospital discharge, and duration of analgesia.

Adverse effects and complications will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Will be included 40 patients, ASA physical status 1 or 2 undergoing hemorrhoidectomy after approval by the Ethics Committee and signed Consent Form.

Exclusion Criteria:

* There will be excluded patients with associated diseases (fistula, fissure) infection at the puncture site, using anticoagulants or analgesics (up to 2 weeks before the procedure) and pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 24 hours
  Numerical score

SECONDARY OUTCOMES:
Time to discharge | 24 hours

OTHER OUTCOMES:
Duration of motor blockade | 24 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borges LA, da Cunha Leal P, Rey Moura EC, Sakata RK. Randomized clinical study on the analgesic effect of local infiltration versus spinal block for hemorrhoidectomy. Sao Paulo Med J. 2017 May-Jun;135(3):247-252. doi: 10.1590/1516-3180.2017.0001260117. Epub 2017 May 29. PMID 28562733